CLINICAL TRIAL: NCT00777751
Title: Radiation Therapy and Cardiac Biomarkers
Brief Title: Radiation Therapy and Cardiac Enzymes
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0489
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Tumor
Keywords: Chest Tumor; Heart; Lung Cancer; Esophageal Cancer; Thymoma; Radiation dose to the heart; Cardiac Enzymes; Cardiac Biomarkers; Radiation Therapy; RT; Electrocardiograms; ECG
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Esophageal Neoplasms; Thymoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this clinical research study is to learn if the radiation that you are receiving will result in an increase in certain proteins produced by the heart called cardiac biomarkers.

DETAILED DESCRIPTION:
Cardiac Biomarkers:

Cardiac biomarkers are proteins made by the heart. When cardiac biomarkers are above normal levels, there may be damage to the heart. The relationship between cardiac biomarkers and radiation therapy has not been well studied. Learning more about this relationship may lead to better ways to check the heart during radiation therapy. How cardiac biomarkers can play a role in predicting future heart problems during radiation therapy will also be studied.

Study Tests:

If you agree to take part in this study, blood (about 1 teaspoon) will be drawn to measure certain cardiac biomarkers up to 2 days before radiation therapy, following the first treatment of radiation, within 2 days of finishing radiation therapy, and about 1 to 2 months after completion of radiation therapy. Once the blood testing is completed, any leftover blood samples will be destroyed.

You will also have electrocardiograms (ECGs -- tests that measure the electrical activity of the heart) at the same time points as the blood draws.

Length of Study:

You will be off study after the last blood draw and ECG.

This is an investigational study. Up to 30 patients will be enrolled in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. A total of thirty patients will be prospectively enrolled in this study. Patients with tumors in the chest including histologically proven primary lung cancer, esophageal cancer, thymoma or mesothelioma to be treated with RT with or without concurrent chemotherapy to a final dose of >/=45 Gy will be included in this study.
2. Patients with tumors in close proximity to the heart where the treating radiation oncologist anticipates the mean cardiac dose will exceed 20Gy.
3. All patients must sign a study-specific informed consent form. If the patient's mental status precludes his/her giving informed consent, written informed consent may be given by the patient's legal representative.
4. Age >/= 18
5. Women of childbearing potential (A woman of child-bearing potential is a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months [i.e., who has had menses at any time in the preceding 24 consecutive months]. For women of childbearing potential, a blood pregnancy test must be performed within 72 hours prior to the start of protocol treatment.

Exclusion Criteria:

1. Patients who receive 5-fluorouracil or adriamycin as part of their chemotherapy regimen.
2. Patients with recent myocardial infarction in the past month, decompensated heart failure or myocarditis/pericarditis in the past month
3. Patients with renal failure indicated by a serum creatinine level of >/= 2.0.
4. Patients in the intensive care unite (ICU).
5. Patients with systemic sepsis.
6. Patients with acute pulmonary embolism in the past month.
7. Women who are pregnant or nursing are not eligible as treatment involves unforeseeable risks to the fetus or child.
8. Inability to obtain histologic proof of malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tumors in the chest in close proximity to the heart, including histologically proven primary lung cancer, esophageal cancer, or thymoma, to be treated with single modality RT.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-10-06 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2016-11-21 (Actual)

PRIMARY OUTCOMES:
Elevation in cardiac biomarkers by measuring cardiac troponins (troponin T and troponin I), BNP, and CK-MB. | 4 Time Points: within 1 week prior to radiation therapy (RT), within 1-3 days of RT completion, and at 1 and 3 months after completion of RT.

CONTACTS AND LOCATIONS:
Overall Officials: David Grosshans, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org